CLINICAL TRIAL: NCT05987046
Title: The Effects of Three Contrast Training Sessions in a Week on Post-activation Countermovement Jump Performance in High Strength Male
Brief Title: Contrast Training, Post-activation Countermovement Jump Performance in High Strength Male
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Tzai-Li Li, Professor, National Taiwan Sport University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NationalTaiwanSportU
Record Dates: First submitted 2023-07-23; First posted 2023-08-14 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast training sessions (Experimental): Participants will perform three contrast training sessions for a week.
  Interventions: Behavioral: Contrast training

INTERVENTIONS:
Behavioral: Contrast training — Three sets of three repetitions of parallel squats at 90% of 1RM

SUMMARY:
The study investigated the effects of three contrast training sessions in a week on post-activation countermovement jump performance in high strength male.

DETAILED DESCRIPTION:
Previous researches indicated that the primary contributor of contrast training to improving explosive performance might be the phenomenon of post-activation performance enhancement (PAPE), with emphasis on conducting plyometric training at the optimal PAPE time. However, the PAPE appeared to be susceptible to fatigue and delayed potentiation of neuromuscular performance. Thus, its applicability in practical training is not yet clarified. The purposes of this study are to: 1) examine the effects of three contrast training sessions in a week on individual and group's PAPE and the optimal timepoint of PAPE; 2) assess the intrasession and intersession reliability of the optimal PAPE timepoints of both individuals and groups; 3) determine the relationship between kinematic parameters during resistance training and PAPE.

Qualified participants will visit the laboratory five times for experimental familiarization, One repetition maximum (1RM) of parallel squat test, and three contrast training sessions, with each contrast training session consisting of three sets of parallel squats in a week. Alongside this, countermovement jump tests will be conducted before the first set of squats and at 1, 3, 5, 7, 9, and 11 minutes after each squat set, with the kinematic parameters of the parallel squats also being collected.

ELIGIBILITY:
Inclusion Criteria:

* Least 2 years of resistance training experience.
* Least 1.75 times body weight of squat 1RM
* Currently engaged in regular exercise training.

Exclusion Criteria:

* Skeletal muscle injury within the past six months.
* Non-responders to PAPE

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
post-activation performance enhancement (PAPE) | Change in baseline and 1, 3, 5, 7, 9, and 11 minutes after each squat set.
  PAPE will be evaluated by maximum height of countermovement jump in this study.
Within-group neuromuscular fatigue | Up to 2 weeks.
  Within-group neuromuscular fatigue will be evaluated by velocity loss rate calculated from maximum and minimum concentric mean velocities of each set for squat in this study.
Between-group neuromuscular fatigue | Up to 2 weeks.
  Between-group neuromuscular fatigue will be evaluated by the fastest mean concentric velocity of each squat set in this study.
Between-day squat performance | Up to 2 weeks.
  Between-day squat performance will be evaluated by the fastest mean concentric velocity of first squat set for each contrast training in this study.
Delayed potentiation of neuromuscular performance (DPNP) | Up to 2 weeks.
  DPNP will be evaluated by maximum height of countermovement jump in this study.

SECONDARY OUTCOMES:
Weight | Baseline
  Weight in kilograms.
Height in meters | Baseline
  Height in meters.
Body fat | Baseline
  The body weight and fat weight will be combined to calculate the body fat in percentage.
Squat 1RM | Baseline
  Squat 1RM will be evaluated maximum weight lifted for 1 repetition of squat in this study.
Concentric mean force of squat | Up to 2 weeks.
  Concentric mean force in newtons.
Concentric peak force of squat | Up to 2 weeks.
  concentric peak force in newtons.
Concentric mean velocity of squat | Up to 2 weeks.
  Concentric mean velocity in meters per second.
Concentric mean velocity loss of squat | Up to 2 weeks.
  Concentric mean velocity loss in percentage.
Concentric peak velocity of squat | Up to 2 weeks.
  Concentric mean velocity in meters per second.
Concentric mean power of squat | Up to 2 weeks.
  concentric mean velocity in watts.
Concentric peak power of squat | Up to 2 weeks.
  Concentric peak power in watts.
Concentric rep duration of squat | Up to 2 weeks.
  Concentric rep duration in scend.
Dip of squat | Up to 2 weeks.
  Dip in meters.
Eccentric min velocity of squat | Up to 2 weeks.
  Eccentric min velocity in meters per second.
Eccentric peak velocity of squat | Up to 2 weeks.
  Eccentric peak velocity in meters per second.
Eccentric peak force of squat | Up to 2 weeks.
  Eccentric peak force in newtons.
Vertical distance of squat | Up to 2 weeks.
  Vertical distance in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Tzai-Li Li, Phd, Study Director — National Taiwan Sport University
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan